CLINICAL TRIAL: NCT07211984
Title: Evaluation of the Clinical and Organizational Impact of the Digital Medical Device Dalia in the Management of Depression
Brief Title: Evaluation of Dalia Solution For Depressed Patient
Acronym: DaliaMonitorin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A01266-43
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Depression Chronic; Depressed; Depressed Mood; Depression and Quality of Life; Depression Diagnosis
Keywords: Depression; PHQ-9; MADRS; Depressive episode; Anxiety disorder; Antidepressant prescriptions; Smartwatch
MeSH Terms: conditions — Consciousness Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients assigned to the "control" group will follow conventional healthcare. According to french "Haute Autorité de Santé", conventional management includes advice on adopting a healthy lifestyle, psychotherapy with a contracted psychologist, and the prescription of antidepressants if necessary. In this case, regular medical follow-up by the general practitioner or psychiatrist is recommended, particularly at the start of antidepressant treatment (notably after the first and second week). Follow-up consultations to assess treatment response should be performed by the physician between M1 and M2, then at M3, M6, and M12, with a frequency adapted according to the clinical evolution of the patient
  Interventions: Other: Conventional healthcare
- Interventional Arm (Experimental): Patients assigned to the "intervention" group will benefit from Dalia telemonitoring in addition to conventional management.
  Interventions: Device: Dalia Monitoring

INTERVENTIONS:
Device: Dalia Monitoring — All patients consulting psychiatrists and general practitioners in participating centers, meeting all eligibility criteria and agreeing to participate in the study, will be consecutively selected and randomized into one of the two groups. For iInterventional arm: Patients will benefit from Dalia telemonitoring, in addition to conventional care.
  Arms: Interventional Arm
Other: Conventional healthcare — All patients consulting psychiatrists and general practitioners in participating centers, meeting all eligibility criteria and agreeing to participate in the study, will be consecutively selected and randomized into one of the two groups. For Control arm: Patients in this group will benefit from the conventional care pathway.
  Arms: Control Group

SUMMARY:
The goal of this superiority clinical investigation, prospective, multicenter, controlled, randomized, open-label is to evaluate the clinical impact of the Dalia medical telemonitoring device on the management of depressive patients. The main question it aims to answer is: the percentage of patients with clinically significant improvement at 3 months. A clinically significant improvement is defined as a decrease of at least 5 points from the initial PHQ-9 score AND/OR a PHQ-9 score lower than 15. The threshold of 5 points is the Minimal Clinically Important Difference (MCID) of the PHQ-9 scale

DETAILED DESCRIPTION:
Worldwide, depression is a disease that affects 3.8% of the population, i.e., about 280 million people [1]. INSERM specifies that major depressive disorder affects all ages of life and concerns about 15 to 20% of the general population [2]. In France, 12.5% of people aged 18-85 years had a history of major depressive episode (MDE) during the past 12 months in 2021 [3]. In 2017, the prevalence of MDE during the past 12 months was 8.2% among the employed French active population [4].

The diagnosis of MDE is clinical. The symptoms of an MDE must persist for at least 2 weeks, and each of them at a certain degree of severity, almost every day. These symptoms must represent a change compared to the patient's usual functioning (professional, social, family) and cause significant distress. Among the main symptoms: depressed mood, loss of interest, dejection, loss of energy, increased fatigability [5]. Standardized assessment tools are diagnostic aids, notably the Patient Health Questionnaire-9 (PHQ-9), the Montgomery-Åsberg Depression Rating Scale (MADRS), the Beck Depression Inventory-II (BDI-II), the Hospital Anxiety and Depression Scale (HADS), and the Hamilton Depression Rating Scale (HDRS) [5].

A first depressive episode may be isolated and resolve spontaneously within six to nine months without specific treatment. However, in most cases, drug treatment is necessary. As a rule, after 8 weeks of a well-conducted drug treatment, one third of patients show complete remission of symptoms, one third show partial remission, and one third do not respond to treatment [2]. One of the main clinical aspects of depression is its recurrent nature. The risk of having another depressive episode gradually increases after each decompensation. Thus, after a first decompensation, more than 50% of individuals will develop a second depressive episode. After two episodes, the relapse rate increases to 70%, and beyond three episodes, to 90% [6].

Due to its consequences at the individual and societal level, depression is a major public health issue, generating high costs related to absenteeism but also to the overall management of affected individuals [7-9]. Indeed, depression impairs the daily functioning, social and professional relationships of affected individuals, and is associated with suicidal behaviors that are very frequent in these individuals. In France, mental health is now a priority, with health insurance expenditures exceeding 23 billion euros in 2023 [8,9]. When including indirect costs, total expenditures related to psychiatric illnesses could exceed 163 billion euros, with depressive and anxiety disorders being among the main causes of years of life lost due to disability [10].

Based on data from the literature, during a major depressive episode, several physical and physiological parameters (heart rate, physical activity, oxygen saturation, and body temperature) are disrupted [13-23]. Continuous monitoring of these parameters would make it possible to better characterize depressive patients and to detect early relapse/recurrence. Early detection of the risk of relapse and recurrence of MDEs could allow for early management.

In France, geographical disparities in the distribution of psychiatrists, with a high concentration in Île-de-France compared to other regions, limit access to care for patients requiring their expertise [22-24]. General practitioners have become the main resource for patients suffering from mental disorders or psychological distress. Indeed, it is estimated that 15 to 40% of the active patient load of general practitioners present a mental disorder or psychological distress [25,26]. However, although trained in the management of somatic pathologies, general practitioners sometimes lack specific skills to recognize, support, and thoroughly treat mental disorders. This often leads to limited management and high prescription of psychotropic drugs. It is estimated that 90% of first-line antidepressant prescriptions come from general practitioners, but follow-up remains insufficient [25,27].

In the literature, digital solutions such as mobile applications have demonstrated their effectiveness in improving mental well-being and reducing symptoms of depression and anxiety [28-31]. Indeed, several systematic reviews and meta-analyses have reported the effectiveness of mHealth interventions based on applications for the management of anxiety and depression symptoms, with effects ranging from small to moderate compared to control groups [32-34]. Medical telemonitoring could play a key role in facilitating this coordination and follow-up of patients by generating alerts adapted to their situation. These data, integrated via dedicated solutions, allow real-time adjustment of the specific management of each patient according to the needs and circumstances generating this alert. However, in France, there is currently no medical telemonitoring device in mental health reimbursed by Health Insurance. Standard follow-up consultations do not always allow continuous monitoring of the patient's condition fluctuations; hence the need for tools enabling early detection of worsening depressive symptoms.

Telemonitoring interventions for depressive patients are generally based on digital tools allowing patients to report their symptoms and health behaviors. This information, called ePROs (electronic Patient-Reported Outcomes), is transmitted to healthcare professionals for continuous monitoring. This approach facilitates the early detection of symptoms, improves communication between patients and caregivers, and allows rapid intervention if necessary. The integration of a telemonitoring solution, Dalia, which continuously collects physiological parameters, offers a considerable advantage compared to a simple collection of ePROs. Indeed, ePROs rely on the patient's subjective reports, which may lead to biases related to the perception or memory of symptoms, and their collection is generally limited to fixed intervals. On the other hand, continuous monitoring of physiological parameters, such as heart rate, oxygen saturation, physical activity, and body temperature, makes it possible to obtain objective and real-time data, thus offering a more complete and accurate picture of the patient's condition. This approach not only allows subtle changes and early signs of worsening to be detected before they are even perceived by the patient, but also to personalize interventions proactively, thus reducing the risks of relapse or hospitalization.

By cross-referencing these physiological data with ePROs, it becomes possible to identify therapeutic needs more quickly and adjust treatment, thereby optimizing depression management and improving long-term outcomes.

We therefore hypothesize that the monitoring of depressive patients through Dalia telemonitoring would improve the response to antidepressant treatment, and reduce the risk of relapse, recurrence, as well as the risk of rehospitalization, emergency room visits, and the number of unscheduled consultations; hence the interest of this clinical investigation evaluating the clinical and organizational impact of the Dalia telemonitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with a diagnosis of depressive episode, as defined by ICD-11, and with a PHQ-9 score ≥ 15 confirmed by a psychiatrist or general practitioner
* Patient receiving a first antidepressant treatment (treatment-naïve) OR having had a modification of antidepressant treatment in the two weeks prior to inclusion
* Patient equipped with a smartphone or a computer or a tablet with internet access
* Patient affiliated to a health insurance scheme
* Patient able to read and understand French
* Patient having signed informed consent

Exclusion Criteria:

* Patient under non-cardioselective beta-blocker (carvedilol, labetalol, propranolol, pindolol) and beta-mimetic (salbutamol, terbutaline)
* Patient with a pacemaker or with a known cardiac arrhythmia
* Patient with major neurocognitive disorder (e.g., dementia) or psychotic disorders likely to compromise participation in the study
* Patient hospitalized at the time of inclusion whose discharge is not planned within the next two weeks
* Patient treated with esketamine
* Patient with excessive consumption of psychoactive substances (alcohol or drugs), which may interfere with the course or follow-up of the study
* Patient unable to wear the bracelet during the study due to dermatological conditions
* Patient under guardianship, curatorship, or legal protection, or any other administrative or judicial measure depriving rights and freedom
* Patient considered non-autonomous by the investigator
* Patient already included in another interventional research study
* Vulnerable persons referred to in Articles L.1121-5 to 8 and L.1122-1-2 of the French Public Health Code are excluded from the study

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months after inclusion
  The primary endpoint will be the percentage of patients with clinically significant improvement at 3 months.
  A clinically significant improvement is defined as a decrease of at least 5 points from the initial PHQ-9 score AND/OR a PHQ-9 score lower than 15.
  The threshold of 5 points is the Minimal Clinically Important Difference (MCID) of the PHQ-9 scale

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Mouchabac, Doctor, Principal Investigator — Dalia Care
Locations (1):
- Neurostim Luxembourg, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor Website — https://www.daliacare.com